CLINICAL TRIAL: NCT00779922
Title: Pharmacokinetics of Lenalidomide (Revlimid®) in Patients With Multiple Myeloma and Impaired Renal Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Frank BRIDOUX - MD - Prof - principal investigator
Other Study IDs: REVIR
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma; Impaired Renal Function
Keywords: Multiple Myeloma; impaired renal function
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 1 to 5 (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profile of Revlimid® in patients presenting with Multiple Myeloma and impaired renal function, the safety of Revlimid® in the enrolled patients population.

and evaluate the efficacy of Revlimid®-Dexamethasone combination in patients presenting MM and impaired renal function at completion of 3 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of relapsed or refractory multiple myeloma (MM).
* Age > 18 years at the time of signing the informed consent form
* Stable renal function

Exclusion Criteria:

* Documented amyloidosis
* Any prior use of Revlimid ®
* Any contraindication to Revlimid ® and especially:
* Lack of acceptable method of birth control for female of childbearing potential (FCPB)

  * Men who don't agree to use condom during the study and 4 weeks after the last study drug intake if their partner is a FCPB.
  * Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France